CLINICAL TRIAL: NCT06901414
Title: Birth Complications and Intrauterine Constraints in the Etiology of Congenital Muscular Torticollis: A Nationwide Registry Study
Status: Completed | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CMT Etiology
Record Dates: First submitted 2025-03-22; First posted 2025-03-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Congenital Muscular Torticollis
Keywords: Congenital muscular torticollis; Birth trauma; crowding; etiology; birth registry
MeSH Terms: conditions — Congenital torticollis; Birth Injuries; Crowding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CMT cases: Children identified in the Norwegian Patient Registry (NPR) with the diagnosis of congenital muscular torticollis (ICD-10 Q68.0) born between 1990 and 2023
- Matched control group: Consisting of individuals from the general population, matched in a 1:4 ratio based on birth year, sex, and gestational age at birth.

SUMMARY:
This retrospective register-based cohort study investigates the association between birth complications, intrauterine crowding, and the development of congenital muscular torticollis (CMT). CMT is characterized by the shortening and tightening of the sternocleidomastoid muscle, leading to abnormal head positioning. The study will analyze data from the Norwegian Medical Birth Registry (MFR) and the Norwegian Patient Registry (NPR) to determine whether individuals with CMT have a higher prevalence of birth complications or signs of intrauterine crowding compared to the general population. By identifying risk factors associated with CMT, this study aims to identify the possible etiology of CMT.

DETAILED DESCRIPTION:
Congenital Muscular Torticollis (CMT) is a condition affecting infants, characterized by a shortened and tightened sternocleidomastoid muscle (SCM), resulting in abnormal head positioning. Despite various theories, the exact etiology of CMT remains unclear. Two primary hypotheses include birth trauma and intrauterine crowding. Some studies have suggested an association between CMT and operative deliveries, whereas others have found no such association. Similarly, intrauterine crowding, such as in multiple pregnancies, has been proposed as a contributing factor due to mechanisms like ischemia or compartment syndrome.

While most children with CMT experience a mild condition that resolves with stretching and physiotherapy, a notable overrepresentation of complicated deliveries has been observed among patients requiring surgical intervention for CMT. This study aims to further explore these hypotheses by analyzing data from the Norwegian Medical Birth Registry (MFR).

Study Objectives The primary objective of this study is to compare the prevalence of operative deliveries and indicators of intrauterine crowding between individuals diagnosed with CMT and the general population. The study seeks to determine whether complicated deliveries and/or crowding are overrepresented among patients with CMT. Specifically, the study will investigate whether there is an increased occurrence of restricted intrauterine conditions or operative deliveries in CMT patients compared to the general birth cohort. If a significant association is found, it would support the hypothesis that these factors contribute to the development of CMT.

Expected Outcomes By conducting this study, we expect to contribute to a better understanding of the potential causes of CMT. The findings may improve early identification and potentially influence obstetric and neonatal management strategies.

Methods This is a registry-based study utilizing anonymized data from the Norwegian Patient Registry (NPR) and linking it to the MFR. The study will identify a cohort of individuals diagnosed with CMT and a matched control group (1:4) from the general population.

Study Design Type: Retrospective, cohort, observational, registry-based study. Matching: Cases will be matched with controls based on birth year, sex, and gestational age at birth in a 1:4 ratio.

Population: Patients diagnosed with CMT who have undergone surgery in Norway, born between 1990 and 2023, will be identified using ICD-10 code Q68.0 and procedure codes NAL39/NAL69/NAL99.

Variables

The study will collect data on variables relevant to birth trauma and crowding hypotheses:

Birth Trauma Indicators:

* Mode of delivery (spontaneous vaginal delivery, assisted vaginal delivery, cesarean section)
* Shoulder dystocia indicators (clavicle fracture, brachial plexus injury)
* Birth weight (>4000g, macrosomia)
* Breech presentation (vaginal delivery)
* Vacuum-assisted delivery
* Forceps-assisted delivery
* Emergency cesarean section due to mechanical complications
* Indications for cesarean section (maternal or fetal factors)

Crowding Indicators:

* Multiple pregnancies (number of fetuses per pregnancy)
* Amniotic fluid levels (normal vs. polyhydramnios)
* Fetal position at birth (cephalic, breech, transverse)
* Birth weight and length relative to gestational age
* Gestational duration (preterm, full-term, post-term)
* Maternal height
* Birth order (firstborn vs. later-born)

Data Collection Data will be retrieved from MFR and NPR through Helsedata.no. The collected data will be anonymized to ensure compliance with ethical guidelines.

Statistical Analysis

The study will employ appropriate statistical methods to compare the prevalence of the examined variables between the CMT cohort and the control group:

* Descriptive statistics to summarize demographic and clinical variables.
* Univariate analysis (Chi-square or Fisher's exact test) to compare the frequency of complicated deliveries between groups.
* Multivariate logistic regression analysis to adjust for confounding variables, including maternal age, comorbidities, gestational age, birth weight, and delivery method.
* Directed Acyclic Graphs (DAGs) will be utilized to illustrate causal relationships.

Limitations

* Potential limitations in available data from MFR.
* Retrospective study design with possible missing or incomplete data.
* The need to differentiate between the causality of crowding and operative delivery, as crowding may necessitate operative delivery.
* Variability in delivery methods across hospitals.
* Selection bias in operative deliveries due to pre-existing intrauterine conditions.

Ethical Considerations Ethical approval will be obtained from the Regional Committees for Medical and Health Research Ethics (REK) and the local privacy protection officer (PVO) at Vestre Viken. The study will use de-identified registry data to maintain participant confidentiality. There will be no direct patient involvement, ensuring compliance with ethical standards.

This study is expected to provide significant insights into the etiology of CMT, contributing to better prevention and management strategies for affected individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with congenital muscular torticollis (ICD-10 code: Q68.0) and registered in the Norwegian Patient Registry (NPR).
* Born in Norway after 1990
* Underwent surgical treatment for CMT (procedure codes NAL39/NAL69/NAL99).

Exclusion Criteria:

* Individuals with incomplete birth registry data in the MFR.
* Presence of congenital anomalies unrelated to CMT that could confound study outcomes.
* Cases with missing gestational age, birth weight, or delivery method.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include a cohort of individuals diagnosed with congenital muscular torticollis (CMT) who have been diagnosed and/or undergone surgical treatment in Norway during the time period of 1990 to 2023. These cases will be identified from the Norwegian Patient Registry (NPR) based on diagnosis and procedure codes. The control group will consist of individuals from the general population, matched in a 1:4 ratio based on birth year, sex, and gestational age at birth. The study will analyze perinatal and birth-related factors, such as mode of delivery, signs of birth trauma, and intrauterine conditions, using data from the Norwegian Medical Birth Registry (MFR).
Sampling Method: Probability Sample
Enrollment: 7105 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Use of vacuum, forceps extraction | Data from the time period of 1990 to 2023.
  The use of vacuum extraction or forceps (operative deliveries), indicates birth complications. It has been hypothesized that such operative deliveries are associated with an increased incidence of congenital muscular torticollis.
  These variables are consistently registered in the Norwegian Birth Registry and have been made accessible to us from the Norwegian Helsedata.no registers.

SECONDARY OUTCOMES:
Caesarean section | 1990-2023
  Caesarean sections will be indentified and compared within groups. One hypothesis is that a caeserian section can protect against CMT by avoiding a possible birth trauma. These variables are consistently registered in the Norwegian Birth Registry and have been made accessible to us from the Norwegian Helsedata.no registers.
Breech position | 1990-2023
  Breech position is possibly associated with both crowding and birth trauma. This variable is consistently registered in the Norwegian Birth Registry and have been made accessible to us from the Norwegian Helsedata.no registers.
Clavicle fracture | 1990-2023
  Clavicle fractures may indicate a birth trauma. These variables are consistently registered in the Norwegian Birth Registry and have been made accessible to us from the Norwegian Helsedata.no registers.
Macrosomic infants | 1990-2023
  Birth weight is routinely registered, with a particular focus on macrosomic infants (>4,000 g birth weight), as it has been hypothesized that macrosomic infants carries a larger risk for CMT (due to the increased risk for a birth trauma).
  This variable is consistently registered in the Norwegian Birth Registry and have been made accessible to us from the Norwegian Helsedata.no registers.
Multiple gestations | 1990-2023
  Multiple gestations, such as twins or higher-order pregnancies, indicate possible crowding. This variable is consistently registered in the Norwegian Birth Registry and have been made accessible to us from the Norwegian Helsedata.no registers.
Amniotic fluid levels | 1990-2023
  Amniotic fluid levels (oligohydramnion/polyhydramnion) may indicate crowding. Crowding har been associated with a higher risk of CMT, causing (possibly) a compartment syndrome within the sternocleid muscles. This variable is consistently registered in the Norwegian Birth Registry and have been made accessible to us from the Norwegian Helsedata.no registers.
Maternal height | 1990-2023
  Maternal height may be associated with increased risk of both crowding and birth complications. This variable is consistently registered in the Norwegian Birth Registry and have been made accessible to us from the Norwegian Helsedata.no registers.

CONTACTS AND LOCATIONS:
Locations (1):
- Vestre Viken HF, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No
Despite the fact that our data are non-identifiable, the permission granted us by the Regional Ethics Committee does not allow us to share data outside our study group.